CLINICAL TRIAL: NCT03516058
Title: Impact Assessment of Simulation-Based Education on Anesthesiology Trainee in Ultrasound-Guided Transversus Abdominis Plane Block Using an Anesthetized Porcine Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4-2018-0208
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Anesthesiology Trainee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Simulation-Based Education — Participating residents receive lectures on TAP block and the use of ultrasound devices from an expert before training, and then receive simulation-based training for an hour from the anesthesiologist's staff. The residents performed three ultrasound guided TAP blocks using an anesthetized porcine model during the training session.
  The residents filled out a questionnaire before and after the training session. Ten multiple-choice questions tested general knowledge in abdomen ultrasound and TAP block. Subjective comfort levels with ultrasound machine and block device functionality, patient positioning, proper block technique, image documentation, needle safety and overall procedural confidence and anxiety levels were reported on a 5-point Likert scale before and after training.

SUMMARY:
The purpose of this study was to investigate the effect of simulation based practice on anesthesiology trainee in ultrasound-guided transversus abdominis plane(TAP) block using an anesthetized porcine model.

The residents filled out a questionnaire before and after the training session. The questionnaires consisted of knowledge including ultrasound anatomy and block technique, comfort, confidence, and axiety levels for the TAP block.

ELIGIBILITY:
Inclusion Criteria:

* Participants included second-year residents, third-year residents who can participate in the anesthesiology simulation training.

Exclusion Criteria:

* None

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
impact of a simulation-based ultrasound-guided TAP block training session_Comfort level | within 1 week after training session
  5-point Likert scale (1 = very low, 2 = low, 3 = moderate, 4 = high, 5 = very high
impact of a simulation-based ultrasound-guided TAP block training session_Comfort level | within 2 months after training session
  5-point Likert scale (1 = very low, 2 = low, 3 = moderate, 4 = high, 5 = very high
impact of a simulation-based ultrasound-guided TAP block training session_Overall confidence level | within 1 week after training session
  5-point Likert scale (1 = very low, 2 = low, 3 = moderate, 4 = high, 5 = very high
impact of a simulation-based ultrasound-guided TAP block training session_Overall confidence level | within 2 months after training session
  5-point Likert scale (1 = very low, 2 = low, 3 = moderate, 4 = high, 5 = very high
impact of a simulation-based ultrasound-guided TAP block training session_Overall anxiety level | within 1 week after training session
  5-point Likert scale (1 = very low, 2 = low, 3 = moderate, 4 = high, 5 = very high
impact of a simulation-based ultrasound-guided TAP block training session_Overall anxiety level | within 2 months after training session
  5-point Likert scale (1 = very low, 2 = low, 3 = moderate, 4 = high, 5 = very high

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine , Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No